CLINICAL TRIAL: NCT06478212
Title: A Phase 1b/2, Multicenter Study of Vorasidenib in Combination With Temozolomide (TMZ) in Participants With IDH1- or IDH2-mutant Glioma
Brief Title: Vorasidenib in Combination With Temozolomide (TMZ) in IDH-mutant Glioma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: S095032-211
Expanded Access: NCT05592743 (Approved for marketing)
Record Dates: First submitted 2024-06-17; First posted 2024-06-27 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: IDH1-mutant Glioma; IDH2-mutant Glioma
Keywords: IDH-mutant glioma; IDH mutation; vorasidenib; S95032; Phase 1/2; pediatric
MeSH Terms: interventions — vorasidenib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1b: Vorasidenib and Temozolomide (TMZ) (Experimental)
  Interventions: Drug: Vorasidenib; Drug: Temozolomide (TMZ)
- Phase 2: Vorasidenib recommended combination dose (RCD) and Temozolomide (TMZ) (Experimental)
  Interventions: Drug: Vorasidenib; Drug: Temozolomide (TMZ)

INTERVENTIONS:
Drug: Vorasidenib — To be taken by mouth once daily in 28-day cycles with no break between cycles
Drug: Temozolomide (TMZ) — To be taken by mouth once daily for the first 5 days of each 28-day cycle, for a maximum of 12 cycles

SUMMARY:
The objective of this study is to determine the safety and tolerability of vorasidenib in combination with temozolomide (TMZ) and to establish the recommended combination dose (RCD) of vorasidenib. The study will begin as a Phase Ib study to determine the RCD and then will transition to a Phase II study to assess the clinical efficacy of vorasidenib at the RCD in combination with TMZ. During the treatment period participants will have study visits on day 1 and 22 of each cycle, with additional visits occurring during the first cycle of the Phase 1b study. Approximately 30 days after treatment has ended, a safety follow-up visit will occur and then participants will be followed for survival every 3 months. Study visits may include questionnaires, blood tests, ECG, vital signs, and a physical examination.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥12 years of age with a weight at screening ≥40 kg.
* Have documented IDH1 or IDH2 mutation based on local testing of tumor tissue by an accredited laboratory
* Have adequate renal function, defined as a creatinine clearance ≥40 mL/min based on the Cockcroft-Gault glomerular filtration rate estimation: (140 - Age) × (Weight in kg) × (0.85 if female) / 72 × serum creatinine (mg/dL).
* Have adequate bone marrow function as evidenced by:

  1. Absolute neutrophil count ≥1,500/mm3 or 1.5×109/L
  2. Hemoglobin ≥9 g/dL or 90 g/L
  3. Platelets ≥100,000/mm3 or 100×109/L
* Have expected survival of ≥3 months.
* KPS or LPPS ≥70 at the start of study treatment.
* Participants on corticosteroids for reasons related to glioma must be on a stable or decreasing dose (≤4mg/day dexamethasone or equivalent) for ≥5 days before the start of study treatment.
* Female participants of reproductive potential must have a negative serum pregnancy test before starting study treatment.

Phase 1b ONLY:

* Have histologically confirmed Grade 2, 3 or 4 IDHm (as per WHO 2021) glioma (astrocytoma or oligodendroglioma).

  1. For oligodendroglioma: Have local testing at an accredited laboratory demonstrating presence of 1p19q co deletion
  2. For astrocytoma: Have local testing by an accredited laboratory demonstrating lack of 1p19q co-deletion and/or documented loss of nuclear ATRX expression or ATRX mutation
* Are appropriate to receive TMZ as post-radiotherapy (RT) adjuvant therapy or as treatment for first disease recurrence after prior RT and/or chemotherapy, per Investigator judgement. For those receiving TMZ in the post-RT adjuvant setting, study treatment must begin no more than 6 weeks after completion of RT.
* Have adequate hepatic function as evidenced by:

  1. Serum total bilirubin ≤1.5×upper limit of normal (ULN); if ≥1.5×ULN and due to Gilbert syndrome, total bilirubin ≤3×ULN with direct bilirubin ≤ULN,
  2. AST and ALT ≤ULN, and
  3. Alkaline phosphatase ≤2.5×ULN.

Phase 2 ONLY:

* Have histologically confirmed Grade 4 astrocytoma, IDHm (per 2021 WHO criteria). Those who meet the Grade 4 designation via homozygous deletion of CDKN2A/B are eligible.
* Have absence of 1p19q co-deletion (i.e., non-co-deleted, or intact) and/or documented loss of nuclear ATRX expression or ATRX mutation by local testing.
* Have received SOC RT with concurrent TMZ (RT-TMZ) before enrollment. Study treatment must begin no more than 6 weeks after completion of RT-TMZ.
* Have adequate hepatic function as evidenced by:

  1. Serum total bilirubin ≤1.5×ULN; if ≥1.5×ULN and due to Gilbert syndrome, total bilirubin ≤3×ULN with direct bilirubin ≤ULN,
  2. AST and ALT at or below the upper limit of normal. An elevation ≤1.5×ULN and considered not clinically significant by the Investigator may be allowed after Medical Monitor (Sponsor) approval, and
  3. Alkaline phosphatase ≤2.5×ULN.

Exclusion Criteria:

* Unable to swallow oral medication.
* Are pregnant or breastfeeding.
* Are participating in another interventional study at the same time; participation in non-interventional registries or epidemiological studies is allowed.
* Have leptomeningeal disease.
* Have a known coagulopathy.
* Received prior therapy with an IDH inhibitor, IDH-directed vaccine, or bevacizumab.
* Have a history of another concurrent primary cancer, with the exception of:

  1. curatively resected non-melanoma skin cancer, or
  2. curatively treated carcinoma in situ. Participants with other previously treated malignancies are eligible provided they have been disease-free for 3 years at Screening.
* Have a known diagnosis of replication repair-deficient glioma (e.g., a known diagnosis of constitutional mismatch repair deficiency or Lynch syndrome).
* Have a known hypersensitivity to any of the components or metabolites of vorasidenib or TMZ.
* Have significant active cardiac disease within 6 months before Screening, including New York Heart Association (NYHA) Class III or IV congestive heart failure, myocardial infarction, unstable angina, and/or stroke.
* Have heart rate corrected QT interval (using Fridericia's formula) (QTcF) ≥450 msec or have other factors that increase risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome). Right bundle branch block and prolonged QTcF interval may be permitted based on local cardiology assessment.
* Have known active hepatitis B (HBV) or hepatitis C (HCV) infections, known positive human immunodeficiency virus (HIV) antibody results, or acquired immunodeficiency syndrome (AIDS) related illness. Participants with a sustained viral response to HCV treatment or immunity to prior HBV infection will be permitted. Participants with chronic HBV or HIV that is adequately suppressed per institutional practice will be permitted.

Phase 1b ONLY:

* For those receiving TMZ in the frontline post-RT adjuvant setting: Have progressive disease during RT or after completion of SOC RT and before the start of study treatment.
* For those receiving TMZ in the recurrent disease setting:

  1. Have received prior systemic anti-cancer therapy (other than surgery) within 1 month (or 6 weeks for nitrosoureas and 6 months for TMZ) of the start of study treatment. In addition, the first dose of study treatment should not occur before a period of 28 days or ≥5 half-lives of any prior investigational agent have elapsed, whichever is longer.
  2. Have received more than one prior line of therapy for glioma (Note: prior RT + chemotherapy is considered one line of therapy).
* Had Grade ≥2 hepatic-related toxicity (AST, ALT, and/or bilirubin elevations) during prior systemic chemotherapy
* Had Grade 4 hematologic toxicity (excluding lymphopenia) that did not recover within 7 days during a prior course of TMZ

Phase 2 ONLY:

* Have received any other glioma-directed therapy other than surgery and SOC RT-TMZ
* Have progressive disease during RT-TMZ or after completion of SOC RT-TMZ and before the start of study treatment.
* Had Grade 4 hematologic toxicity (excluding lymphopenia) that did not recover within 7 days during concurrent RT-TMZ
* Had Grade ≥2 hepatic-related toxicity (AST, ALT, and/or bilirubin elevations) during concurrent RT-TMZ

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2025-01-22 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1b ONLY: Dose-limiting toxicities (DLTs) | Through cycle 1 (each cycle is 28 days)
Number and severity of adverse events (AEs), serious adverse events (SAEs), and AEs of special interest (AESIs) | Through 30 days after the end of treatment (Approximately 3 years)
Progression-free Survival (PFS) status at 12 months | 12 months after treatment initiation

SECONDARY OUTCOMES:
PFS | Through study completion (Approximately 3 years)
Overall survival (OS) | Through study completion (Approximately 3 years)
Objective response rate (ORR) | Through study completion (Approximately 3 years)
Clinical benefit rate (CBR) (CR+partial response [PR]+stable disease [SD]) | Through study completion (Approximately 3 years)
Plasma concentration of vorasidenib and its metabolite AGI-69460 | Through cycle 13 (each cycle is 28 days)
Phase 1b ONLY: Plasma concentration of TMZ | Through cycle 2 (each cycle is 28 days)
Area under the curve (AUC) of vorasidenib and its metabolite AGI-69460 | Through cycle 13 (each cycle is 28 days)
Time to maximum concentration (Tmax) of vorasidenib and its metabolite AGI-69460 | Through cycle 13 (each cycle is 28 days)
Maximum concentration (Cmax) of vorasidenib and its metabolite AGI-69460 | Through cycle 13 (each cycle is 28 days)
Trough concentration (Ctrough) of vorasidenib and its metabolite AGI-69460 | Through cycle 13 (each cycle is 28 days)
Phase 1b ONLY: Area under the curve (AUC) of TMZ | Through cycle 2 (each cycle is 28 days)
Phase 1b ONLY: Time to maximum concentration (Tmax) of TMZ | Through cycle 2 (each cycle is 28 days)
Phase 1b ONLY: Maximum concentration (Cmax) of TMZ | Through cycle 2 (each cycle is 28 days)
Phase 1b ONLY: Trough concentration (Ctrough) of TMZ | Through cycle 2 (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (6):
  - University of California Los Angeles, Los Angeles, California
  - University of Miami, Miami, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - MD Anderson Cancer Center, Houston, Texas
- Medical University of Vienna - AKH, Vienna, Austria
- China (2):
  - Beijing Tiantan Hospital, Capital Medical University, Beijing
  - Huashan Hospital, Fudan University, Shanghai
- France (3):
  - Hôpital Pierre Wertheimer, Lyon
  - Hôpital Pitié-Salpêtrière, Paris
  - IUCT-Oncopole Institut Universitaire du Cancer, Toulouse
- Germany (3):
  - Universitätsklinikum Heidelberg, Heidelberg
  - Medizinische Fakultät Mannheim, Universität Heidelberg, Mannheim
  - Universitätsklinikum Regensburg, Regensburg
- The Tel Aviv Sourasky Medical Center (TASMC) (Ichilov Hospital), Tel Aviv, Israel
- Italy (3):
  - Instituto Clinico Humanitas IRCCS, Rozzano, Milan
  - IOV - Ospedale Busonera, Padua
  - Ospedale Molinette - Centro Oncologico Ematologico, Turin
- Japan (4):
  - Kumamoto University Hospital, Kumamoto
  - Kyoto University Hospital, Kyoto
  - Nagoya University Hospital, Nagoya
  - National Cancer Center Hospital, Tokyo
- Erasmus MC, Rotterdam, Netherlands
- Spain (2):
  - H. Valle de Hebron, Barcelona
  - Hospital 12 de Octubre, Madrid
- United Kingdom (2):
  - Christie Hospital, Manchester
  - The Royal Marsden in Sutton, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data. Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorization in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com/